CLINICAL TRIAL: NCT00836953
Title: A Trial for the Collection of Sera in Healthy Children Receiving Influenza Virus Vaccine USP Trivalent Types A and B (Zonal Purified Subvirion) Fluzone® 2003/2004
Brief Title: Study to Collect Sera for Immunogenicity Testing in Children Vaccinated With Fluzone®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GRC17
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Results first posted 2009-08-27 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Influenza
Keywords: Influenza; Fluzone®; Children
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Group (Experimental): Participants received 2 doses of Fluzone® vaccine
  Interventions: Biological: Influenza virus vaccine (Pediatric formulation)

INTERVENTIONS:
Biological: Influenza virus vaccine (Pediatric formulation) — 0.25 mL, Intramuscular
  Other Names: Fluzone®

SUMMARY:
To describe the safety findings from Days 0 to 44 following injection of the 2003-2004 pediatric formulation of the inactivated, split-virion influenza vaccine Fluzone®, given in the two-dose schedule in accordance with the Package Insert, in children aged ≥ 6 months to < 36 months.

To describe the immunogenicity findings from Days 0 to 44 following injection of the 2003-2004 pediatric formulation of the inactivated, split-virion influenza vaccine Fluzone®, given in the two-dose schedule in accordance with the Package Insert, in children aged ≥ 6 months to < 36 months

DETAILED DESCRIPTION:
The study is to collect sera from healthy children being administered the 2003-2004 formulation of the inactivated, split-virion influenza vaccine Fluzone®.

ELIGIBILITY:
Inclusion Criteria :

* Aged ≥ 6 months to < 36 months.
* Considered to be in good health on the basis of reported medical history and limited physical examination.
* Available for the duration of the study (44 days +4 days).
* Parent/guardian is willing and able to provide informed consent.
* Parent/guardian is willing and able to meet protocol requirements.

Exclusion Criteria :

* Reported allergy to egg proteins, chicken proteins, or any other constituent of the vaccine.
* Previous history of influenza vaccination or documented history of influenza infection.
* An acute illness with or without fever (temperature > 100.4 °F rectal) in the 72 hours preceding enrollment in the trial (defer enrollment).
* Clinically significant findings in vital signs or review of systems (investigator judgment; defer or exclude).
* Participation in any other clinical trial within 30 days prior to enrollment up to termination of the subject's participation in the study.
* Known or suspected impairment of immunologic function, or receipt of immunosuppressive therapy or immunoglobulin since birth.
* Personal or immediate family history of congenital immune deficiency.
* Developmental delay, neurologic disorder, or seizure disorder.
* Chronic medical, congenital, or developmental disorder.
* Known human immunodeficiency virus (HIV)-positive mother.
* Prior history of Guillain-Barré syndrome.
* Any condition which, in the opinion of the investigator, would pose a health risk to the subject or interfere with the evaluation of the vaccine.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2003-09; Primary Completion 2004-01 (Actual); Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Norfolk, Virginia, United States

REFERENCES:
- [Result] Mitchell DK, Ruben FL, Gravenstein S. Immunogenicity and safety of inactivated influenza virus vaccine in young children in 2003-2004. Pediatr Infect Dis J. 2005 Oct;24(10):925-7. doi: 10.1097/01.inf.0000180978.66362.d9. PMID 16220095
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 11 through 25 September 2003 in 1 US site.
Pre-assignment Details: A total of 33 participants who met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- Study Group: Participants received study vaccine on Days 0 and 30.
Period: Overall Study
Arm/Group | Study Group
Started | 33
Completed | 31
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 33
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Months]
  Age Continuous | 19.08 (9.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Solicited Local and Systemic Reactions After Fluzone® Vaccination
Description: Solicited local reactions: Erythema (redness), induration, bruising and pain at the injection site. Solicited systemic reactions: Fever (temperature), irritability, crying, lethargy, appetite decreased, diarrhea, vomiting and rash.
Time Frame: Day 0 to 3 post-vaccination
Population: Safety analysis was on all enrolled and vaccinated subjects with available reaction data, intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 33
Participants
  Any Solicited Local Reaction Post-Dose 1 | 9
  Any Redness (> 5 mm) | 6
  Grade 3 Redness (> 50 mm) | 0
  Any Induration (> 5 mm) | 2
  Grade 3 Induration (> 50 mm) | 0
  Any Bruising (> 5 mm) | 3
  Grade 3 Bruising (> 50 mm) | 0
  Any Pain | 7
  Grade 3 Pain (Cries when leg or arm is moved) | 0
  Any Solicited Local Reaction Post-Dose 2 | 12
  Any Redness (> 5 mm) | 6
  Grade 3 Redness (> 50 mm) | 0
  Any Induration (> 5 mm) | 5
  Grade 3 Induration (> 50 mm) | 0
  Any Bruising (> 5 mm) | 2
  Grade 3 Bruising (> 50 mm) | 0
  Any Pain | 9
  Grade 3 Pain (Cries when leg or arm is moved) | 0
  Any Solicited Local Reaction Post-Any Dose | 14
  Any Redness (> 5 mm) | 8
  Grade 3 Redness (> 50 mm) | 0
  Any Induration (> 5 mm) | 5
  Grade 3 Induration (> 50 mm) | 0
  Any Bruising (> 5 mm) | 5
  Grade 3 Bruising (> 50 mm) | 0
  Any Pain | 10
  Grade 3 Pain (Cries when leg or arm is moved) | 0
  Any Solicited Systemic Reaction Post-Dose 1 | 19
  Fever (Rectal Temp) | 6
  Grade 3 Fever (> 103.1 ºF) | 2
  Any Irritability | 10
  Grade 3 Irritability (> 3 hours) | 2
  Any Crying | 11
  Grade 3 Crying (inconsolable for > 3 hours) | 1
  Any Lethargy | 9
  Grade 3 Lethargy (Uninterested in usual activity) | 0
  Any Appetite Decreased | 11
  Grade 3 Appetite Decreased (Refuses ≥ 3 feeds) | 1
  Any Vomiting | 3
  Grade 3 Vomiting ( ≥ 3 episodes) | 1
  Any Diarrhea | 6
  Grade 3 Diarrhea ( > 5 diarrhea stools/day) | 0
  Rash - Presence of Welts | 0
  Any Solicited Systemic Reaction Post-Dose 2 | 14
  Fever (Rectal Temp) | 2
  Grade 3 Fever (> 103.1 ºF) | 0
  Any Irritability | 12
  Grade 3 Irritability (> 3 hours) | 0
  Any Crying | 7
  Grade 3 Crying (inconsolable for > 3 hours) | 0
  Any Lethargy | 7
  Grade 3 Lethargy (Uninterested in usual activity) | 0
  Any Appetite Decreased | 8
  Grade 3 Appetite Decreased (Refuses ≥ 3 feeds) | 0
  Any Vomiting | 3
  Grade 3 Vomiting ( ≥ 3 episodes) | 0
  Any Diarrhea | 4
  Grade 3 Diarrhea (> 5 diarrhea stools/day) | 0
  Rash - Presence of Welts | 1
  Any Solicited Systemic Reaction Post-Any Dose | 22
  Any Fever | 7
  Grade 3 Fever (> 103.1 ºF) | 2
  Any Irritability | 15
  Grade 3 Irritability (> 3 hours) | 2
  Any Crying | 12
  Grade 3 Crying (inconsolable for > 3 hours) | 1
  Any Lethargy | 11
  Grade 3 Lethargy (Uninterested in usual activity) | 0
  Any Appetite Decreased | 14
  Grade 3 Appetite Decreased (Refuses ≥ 3 feeds) | 1
  Any Vomiting | 4
  Grade 3 Vomiting (≥ 3 episodes) | 1
  Any Diarrhea | 7
  Grade 3 Diarrhea (> 5 diarrhea stools/day) | 0
  Rash - Presence of Welts | 1

2. Other Pre Specified Outcome: Percentage of Participants With Pre- and Post-Vaccination Reciprocal Hemagglutination Inhibition Titers ≥ 40 (Seroprotection)
Description: Seroprotection defined as percentage of participants with reciprocal hemagglutination inhibition titers ≥40 pre- and post-vaccination.
Time Frame: Day 0 and Day 14 after Dose 2
Population: Immunogenicity analysis was on all enrolled and vaccinated subjects with adequate sera for testing, per-protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Study Group
Number analyzed (Participants) | 31
Percentage of Participants
  A/Panama (H3N2) Pre-vaccination | 10
  A/Panama (H3N2) Post-dose 2 | 77
  A/New Caledonia (H1N1) Pre-vaccination | 10
  A/New Caledonia (H1N1) Post-dose 2 | 81
  B/Hong Kong Pre-vaccination | 0
  B/Hong Kong Post-dose 2 | 48

3. Other Pre Specified Outcome: Percentage of Participants With at Least a 4-fold Rise in Reciprocal Hemagglutination Inhibition Titers (Seroconversion)
Description: Seroconversion defined as the percentage of participants with ≥ 4-fold increases in reciprocal hemagglutination inhibition titer from pre- to post-vaccination.
Time Frame: Day 0 and Day 14 Post-dose 2
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Study Group
Number analyzed (Participants) | 31
Percentage of Participants
  A/Panama (H3N2) | 84
  A/New Caledonia (H1N1) | 94
  B/Hong Kong | 81

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the entire study period, from the day of vaccination to Day 44 post-vaccination.
Arm/Group | Study Group
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 19/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=33)
Constipation (Gastrointestinal disorders) | 2 (2)
Teething (Gastrointestinal disorders) | 2 (2)
Vomiting NOS (Gastrointestinal disorders) | 4 (4)
Pyrexia (General disorders) | 5 (5)
Nasopharyngitis (Infections and infestations) | 9 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications